CLINICAL TRIAL: NCT07038577
Title: Impact of Fenugreek Supplementation on Obesity and Hyperglycemia Among Diabetic Adults in Saudi Arabia: A Quasi-Experimental Study
Brief Title: Impact of Fenugreek Supplementation on Obesity and Hyperglycemia Among Diabetic Adults in Saudi Arabia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hail (Other)
Responsible Party: Principal Investigator, Bushra Alshammari, DR, University of Hail
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UOHail
Record Dates: First submitted 2025-06-09; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Type 2 Diabetes Mellitus (T2DM); Obesity and Type 2 Diabetes; Hyperglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Hyperglycemia

STUDY DESIGN:
Intervention Model Description: Participants were assigned to one of two parallel groups. One group received Fenugreek seed powder along with standard diabetes treatment, while the other group received standard treatment only. Each participant remained in their assigned group for the full duration of the 3-month study period, with no crossover between groups.
Masking Description: All participants, care providers, and investigators were aware of the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Fenugreek Supplementation (Experimental): 40 Participants in this group received 10 grams of Fenugreek seed powder twice daily (before breakfast and dinner) for 3 months, in addition to their usual diabetes treatment and a standard meal plan.
  Interventions: Other: Fenugreek Seed Powder
- Arm 2: Standard Care Only (No Intervention): 40 Participants in this group continued their usual diabetes treatment and followed a standard meal plan. They did not receive the Fenugreek supplement.

INTERVENTIONS:
Other: Fenugreek Seed Powder — Participants in the intervention group received 10 grams of ground Fenugreek seed powder, administered twice daily (before breakfast and dinner), for a total of 3 months. The Fenugreek powder was consumed mixed with water, in addition to the participants' regular antidiabetic medications and a standardized meal plan. The supplement was provided in a non-encapsulated, natural powdered form, and was not combined with any other herbal or pharmaceutical products.
  Arms: Arm 1: Fenugreek Supplementation

SUMMARY:
The goal of this clinical trial is to learn if Fenugreek seed powder helps lower body weight and blood sugar in adults with type 2 diabetes who are overweight or obese. The main questions it aims to answer are:

Does Fenugreek lower body mass index (BMI)? Does Fenugreek lower fasting blood sugar, random blood sugar, and HbA1c levels? Researchers will compare people who take Fenugreek along with their regular diabetes care to people who receive only standard diabetes care, to see if the Fenugreek supplement adds extra benefits.

Participants will:

Take 10 grams of Fenugreek seed powder twice a day (before breakfast and dinner) for 3 months.

Follow their usual diabetes treatment and a recommended meal plan. Visit the clinic four times during the study to check weight and blood sugar levels.

This study is being done in Hail City, Saudi Arabia.

DETAILED DESCRIPTION:
This clinical trial tested whether Fenugreek seed powder, a natural dietary supplement, could help lower blood sugar and reduce body weight in adults with type 2 diabetes. The study was conducted in Hail City, Saudi Arabia, and involved 80 participants who were either overweight or obese and diagnosed with type 2 diabetes.

Participants were assigned to one of two groups:

The intervention group received 10 grams of Fenugreek seed powder twice daily (before breakfast and dinner) for three months, in addition to their usual diabetes treatment and a standard meal plan.

The control group received only their standard diabetes care and meal plan, without the Fenugreek supplement.

The study used a quasi-experimental pretest-posttest design. Participants' weight (BMI), fasting blood sugar (FBS), random blood sugar (RBS), and HbA1c were measured at the start and monitored throughout the three-month period. Data were collected from local clinics and hospitals that serve people with diabetes in the region.

This study aims to provide evidence on the potential role of Fenugreek as a safe, culturally accepted, and cost-effective supplement that can support diabetes management and reduce obesity-related complications in the Saudi population

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18 years or older

Diagnosed with type 2 diabetes mellitus

Body Mass Index (BMI) classified as overweight or obese

Receiving standard diabetes treatment (e.g., oral hypoglycemic agents)

Able and willing to provide informed consent

Residing in Hail City, Saudi Arabia

Exclusion Criteria:

Diagnosed with type 1 diabetes mellitus

Currently using insulin therapy

Pregnant or breastfeeding women

Known allergy or sensitivity to Fenugreek

Diagnosed gastrointestinal diseases or malabsorption conditions

Participation in another clinical trial within the past 3 months

Any serious medical or psychiatric condition that, in the opinion of the investigators, could interfere with study participation

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Change in Body Mass Index (BMI) | Baseline and 3 months after intervention
  BMI will be calculated as weight in kilograms divided by the square of height in meters (kg/m²).

SECONDARY OUTCOMES:
Change in Fasting Blood Sugar (FBS) | Baseline and 3 months after intervention
  Fasting blood sugar will be measured in mg/dL to assess glycemic control
Change in Random Blood Sugar (RBS) | Baseline and 3 months after intervention
  Random blood sugar will be measured in mg/dL to evaluate fluctuations in blood glucose levels.
Change in Hemoglobin A1c (HbA1c) | Baseline and 3 months after intervention
  HbA1c will be measured as a percentage to assess long-term glycemic control.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hail, Hail, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data (IPD) with other researchers.
  The data collected will be used solely for the purposes outlined in the approved research protocol and will remain confidential.
  Any future data sharing (if considered) would require additional ethical clearance and participant consent.

REFERENCES:
- [Result] Neelakantan N, Narayanan M, de Souza RJ, van Dam RM. Effect of fenugreek (Trigonella foenum-graecum L.) intake on glycemia: a meta-analysis of clinical trials. Nutr J. 2014 Jan 18;13:7. doi: 10.1186/1475-2891-13-7. PMID 24438170
- See also: Related Info — https://pmc.ncbi.nlm.nih.gov/articles/PMC11403534/?utm_source=chatgpt.comhttps://pmc.ncbi.nlm.nih.gov/articles/PMC10531284/?utm_source=chatgpt.com

DOCUMENTS (1):
  • Study Protocol (2025-06-10): https://cdn.clinicaltrials.gov/large-docs/77/NCT07038577/Prot_000.pdf